CLINICAL TRIAL: NCT00904566
Title: Validation 70-gene MammaPrint Profile in Japanese Population
Brief Title: Validation of 70-gene MammaPrint Profile in Japanese Population
Status: Completed | Type: Observational
Sponsor: Agendia (Industry)
Collaborators: Osaka General Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MP-107-RR
Record Dates: First submitted 2009-05-18; First posted 2009-05-19 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Breast Cancer
Keywords: microarray; gene expression profiling; MammaPrint; breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
By using gene-expression profiling, Van't Veer and colleagues developed a 70-gene prognosis profile, MammaPrint, to identify breast cancer patients who are at low risk of developing distant metastases and therefore might safely be spared chemotherapy. The aim of this study is to evaluate the prognostic value of the 70-gene Mammaprint profile in Japanese women with node-negative breast cancer.

DETAILED DESCRIPTION:
Frozen tumor samples from 140 node-negative, breast cancer patients aged between 29 and 70 years at diagnosis are hybridized on MammaPrint array. Patients were treated with breast conserving therapy or mastectomy with axillary lymph node dissection between December 1998 and August 2001 at Osaka Medical Center for Cancer and Cardiovascular Diseases. Samples are evaluated by gene expression profiling for the 70-gene MammaPrint profile and classified as genomic high risk or genomic low risk.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients
* Node-negative
* Treated with breast conserving therapy or mastectomy with axillary lymph node dissection at Osaka Medical Center for Cancer and Cardiovascular Diseases

Ages: 29 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients, node-negative, treated with breast conserving therapy or mastectomy with axilary lymph node dissection at Osaka Medical Center for Cancer and Cardiovascular Diseases.
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2008-04; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
The probability of recurrence free survival (PRFS) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Kikuya Kato, MD, PhD, Prof, Study Chair — Osaka Medical Center for Cancer and Cardiovascular Diseases
Locations (1):
- Osaka Medical Center for Cancer and Cadiovascular Diseases, Osaka, Japan

REFERENCES:
- See also: Related Info — http://www.agendia.com